CLINICAL TRIAL: NCT02561845
Title: Effectiveness of Statins on Lipid Goal Attainment and Lipid Parameters in Percutaneous Coronary Intervention Patients
Brief Title: Effectiveness of Statins on Lipid Goal Attainment and Lipid Parameters in PCI Patients
Status: Withdrawn | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3560R00019
Record Dates: First submitted 2015-09-16; First posted 2015-09-28 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: PCI Patients
Keywords: Effectiveness of statins, on lipid goal attainment and lipid parameters in Percutaneous Coronary Intervention patients
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rosuvastatin group: patients who received rosuvastatin
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — 5mg, 10mg, 20mg

SUMMARY:
Most PCI patients are at very high cardiovascular (CV) risk, and as such here is an increased need for intensive lipid management in Percutaneous Coronary Intervention (PCI) patients and the population is well suited to demonstrating rosuvastatin's low density lipoprotein-cholesterol (LDL-C) lowering efficacy.Most PCI patients are at very high CV risk, and as such here is an increased need for intensive lipid management in PCI patients and the population is well suited to demonstrating rosuvastatin's LDL-C lowering efficacy.The purpose of this study is to observe the effectiveness of statins on lipid level reduction (LDL-C, high density lipoprotein-cholesterol (HDL-C), Triglyceride (TG), and non-HDL-C) and lipid goal attainment according to recent guidelines.

DETAILED DESCRIPTION:
The number of patients receiving Percutaneous Coronary Intervention (PCI) is rapidly increasing in China. In 2013, about 450,000 Chinese patients received PCI, most of whom suffered from coronary heart disease (CHD), especially acute coronary syndrome (ACS). ACS is associated with an increased risk of cardiovascular mortality and recurrent cardiac events, underscoring the importance of identifying treatments that minimize this risk.The Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering (MIRACL) trial suggested a benefit of lipid lowering with high-dose atorvastatin in patients with ACS. A meta-analysis of statin use in patients with ACS confirmed the benefits of early high-dose statin administration in decreasing recurrent myocardial ischemia, which suggested the clinical benefit and safety of statins were dose and statin dependent. The updated National Cholesterol Education Program Adult Treatment Panel III guidelines recommend that intensive therapy should be considered for all patients admitted to hospital for an ACS. Two meta-analyses have shown that early intensive statin therapy in patients with ACS is associated with a reduced rate of death and cardiovascular events. In the PROVE IT study, comparing atorvastatin 80 mg with pravastatin 40 mg, a significant reduction in major adverse clinical events was observed in favour of more intensive statin treatment. In that study, the median concentration of low-density LDL-C was lowered from 106 mg/dL to 62 mg/dL in the atorvastatin 80 mg group. More recently, the 2011 European Society of Cardiology (ESC)/ European Arterial Sclerosis Association (EAS) guideline for the management of dyslipidemia recommended patients with ACS are very high CV risk patients and should achieve LDL-C level <70 mg/dl or 50% reduction. In 2011 American College of Cardiology Foundation (ACCF) / American Heart Association (AHA) / (cardiovascular angiography and intervention Association)/ Association of Cardiovascular angiography and intervention (SCAI) Guideline for PCI, statin therapy which lowers LDL to <70mg/dL in very high-risk patients is recommended (IIa, B). The latest China ACS consensus also recommends using the highest dose statin treatment for the acute phase and to attain an LDL-C level of 1.8 mmol/L or 50% reduction compared with baseline in long-term treatment. However, there are very limited Chinese data demonstrating the current situation of lipid management (LDL-C on-goal rate) by different statins in real-world clinical practice.

Most PCI patients are at very high CV risk, and as such here is an increased need for intensive lipid management in PCI patients and the population is well suited to demonstrating rosuvastatin's LDL-C lowering efficacy.Most PCI patients are at very high CV risk, and as such here is an increased need for intensive lipid management in PCI patients and the population is well suited to demonstrating rosuvastatin's LDL-C lowering efficacy.The purpose of this study is to observe the effectiveness of statins on lipid level reduction (LDL-C, HDL-C, TG, and non-HDL-C) and lipid goal attainment according to recent guidelines.

ELIGIBILITY:
Inclusion criteria:

* Patients must have had at least one treatment for statins, during the intake period (between 01/07/2011 and 31/01/2015). The date treated with statins after hospitalization before PCI or after PCI for statin naive patients, and date of PCI procedure for statin users will be marked as an index date.
* Patients must be 18 years or older at the time of index date.
* Patients must have at least 1 month of follow-up after the index date, including continuous statin treatment, lipid profile and lab values for safety profile.
* Patients must have at least two lab values: one full lipid panel prior to or on the index date, and one at least 30 days following the index date.

Exclusion criteria:

* Patients with a diagnosis of Familial Hypercholesterolemia.
* Patients with malignant tumor at the index day.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PCI Patients initiating statin therapy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Low density lipoprotein-cholesterol (LDL-C) at 30 days | Blood samples are collected pre-dose, 30 days post dose
  by assessment of statins on the on-goal rate of LDL-C treatment of patients underwent PCI

SECONDARY OUTCOMES:
Change from baseline lipid level at 30 days | Blood samples are collected pre-dose, 30 days post dose
  by assessment of other lipid level reduction from baseline lab value to the last lab value
Change from baseline lipid level at 3 months | Blood samples are collected pre-dose, 3 months post dose
  by assessment of other lipid level reduction from baseline lab value to the last lab value
Change from baseline lipid level at 6 months | Blood samples are collected pre-dose, 6 months post dose
  by assessment of other lipid level reduction from baseline lab value to the last lab value
Change from baseline lipid level at 12 months | Blood samples are collected pre-dose, 12 months post dose
  by assessment of other lipid level reduction from baseline lab value to the last lab value
number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 at 30 days | Blood samples are collected at 30 days post dose
  by assessment of safety profile
number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 at 3 months | Blood samples are collected at 3 months post dose
  by assessment of safety profile
number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 at 6 months | Blood samples are collected at 6 months post dose
  by assessment of safety profile
number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 at 12 months | Blood samples are collected at 12 months post dose
  by assessment of safety profile
Change from the baseline statin dose at 12 months | The dose of the treated statin is collected up to 12 months
  by assessment of treatment patterns and adherence of the index statin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD,PhD, Principal Investigator — Chinese PLA General Hospital